CLINICAL TRIAL: NCT05692115
Title: Ischemia and Inflammatory Markers Among Patients With Coronary Artery Ectasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Nageh Nanoush Hakeem, Resident, Assiut University
Other Study IDs: Stress ECG,inflammation in CAE
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Ectasia
Keywords: stress ECG and inflammatory markers in Coronary Artery Ectasia
MeSH Terms: conditions — Coronary Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: Coronary Artery Ectasia patients
  Interventions: Diagnostic Test: stress ECG
- control: Normal coronary artery patients
  Interventions: Diagnostic Test: stress ECG

INTERVENTIONS:
Diagnostic Test: stress ECG — stress ECG to patients suspected to be ischemic patients .

SUMMARY:
study the ischemic burden in patients with CAE, and its relation to inflammatory markers.

* To assess the ischemic response during exercise ECG among patients with different variants of CAE.
* To assess inflammatory biomarkers among patient with different variants of CAE
* To assess the relation between the ischemic response and inflammatory markers.

DETAILED DESCRIPTION:
Coronary artery ectasia (CAE) is a dilation of the coronary artery lumen. The term "ectasia" refers to diffuse dilation of a coronary artery, while focal coronary dilation is called a "coronary aneurysm." The definition of coronary artery ectasia is a dilatation exceeding more than one-third of the coronary artery length with the diameter of the dilated segment measuring more than 1.5 times the diameter of a normal adjacent segment. Coronary artery ectasia is well recognized, but uncommon findings encountered during diagnostic coronary angiography.

inflammation, platelet activation, endothelial dysfunction, microvascular dysfunction, slow flow and vascular remodeling have all been suggested to play a role .

. Available evidence implies that CAE is not a mere variant of CAD; indeed diabetes is negatively associated with CAE and studies pinpoint a critical inflammatory component

Turbulent slow flow within dilated coronaries may lead to platelet activation, thrombosis and eventually acute coronary syndrome Local coronary flow disturbances caused by decreased endothelial shear stress has also been proposed as an alternative explanation for the coexistence of CAD and CAE. Intravascular ultrasound (IVUS) evidence suggests that atherosclerotic plaques within ectatic regions of vessels are highly inflamed and meet high-risk plaque criteria

Mediators of chronic inflammation, such as growth factors and cellular adhesion models, have been widely described in the pathogenesis of CAE. Specifically, the expression of specific inflammatory markers, particularly IL-6 and CRP, is known to be higher in CAE compared with CAD and healthy controls . Most recently, a large meta-analysis elucidated the role of other contributory markers, neutrophil to lymphocyte ratio (NLR) and red cell distribution width (RDW), in the pathogenesis of CAE

Inflammatory markers, C-reactive protein and albumin are believed to be involved in the progression and severity of CAE. Recently, a significantly higher C-reactive protein-to-albumin ratio has been associated with isolated CAE when compared to obstructive CAD and controls. Notably, C-reactive protein-to-albumin ratio also correlated strongly with the severity of CAE, which provides further evidence for its potential role in detection and management

We sought to study the ischemic burden in patients with CAE, and its relation to inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with suspected CAD who are undergoing elective coronary angiography.

Exclusion Criteria:

Patients with a history of cardiomyopathy or myocardial infarction (MI). Patients with recent acute coronary syndrome Patients with severe renal impairment Post CABG patients Patients with physical incapacity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cases : Coronary Artery Ectasia patients controls : Normal coronary artery patients
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Ischemia and Inflammatory markers among patients with coronary artery ectasia . | 2 years
  Incidence of exercise induced ischemic changes on stress ECG: ST-T changes and chest pain reported by patient.

SECONDARY OUTCOMES:
Ischemia and Inflammatory markers among patients with coronary artery ectasia . | 2 years
  Assays of inflammatory markers measured at a fixed time interval among patients as: NLR, RDW, hs-CRP, IL6.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mavrogeni S. Coronary artery ectasia: from diagnosis to treatment. Hellenic J Cardiol. 2010 Mar-Apr;51(2):158-63. No abstract available. PMID 20378518
- [Background] Aboeata AS, Sontineni SP, Alla VM, Esterbrooks DJ. Coronary artery ectasia: current concepts and interventions. Front Biosci (Elite Ed). 2012 Jan 1;4(1):300-10. doi: 10.2741/377. PMID 22201872
- [Background] Eitan A, Roguin A. Coronary artery ectasia: new insights into pathophysiology, diagnosis, and treatment. Coron Artery Dis. 2016 Aug;27(5):420-8. doi: 10.1097/MCA.0000000000000379. PMID 27218145
- [Background] Devabhaktuni S, Mercedes A, Diep J, Ahsan C. Coronary Artery Ectasia-A Review of Current Literature. Curr Cardiol Rev. 2016;12(4):318-323. doi: 10.2174/1573403x12666160504100159. PMID 27142049
- [Background] Huang QJ, Liu J, Chen MH, Li JJ. Relation of diabetes to coronary artery ectasia: A meta-analysis study. Anadolu Kardiyol Derg. 2014 Jun;14(4):322-7. doi: 10.5152/akd.2014.5327. Epub 2014 May 2. PMID 24818774
- [Background] Antoniadis AP, Chatzizisis YS, Giannoglou GD. Pathogenetic mechanisms of coronary ectasia. Int J Cardiol. 2008 Nov 28;130(3):335-43. doi: 10.1016/j.ijcard.2008.05.071. Epub 2008 Aug 9. PMID 18694609
- [Background] Dereli S, Cerik IB, Kaya A, Bektas O. Assessment of the Relationship Between C-Reactive Protein-to-Albumin Ratio and the Presence and Severity of Isolated Coronary Artery Ectasia. Angiology. 2020 Oct;71(9):840-846. doi: 10.1177/0003319720930983. Epub 2020 Jun 10. PMID 32519552
- [Background] Shao Q, Chen K, Rha SW, Lim HE, Li G, Liu T. Usefulness of Neutrophil/Lymphocyte Ratio as a Predictor of Atrial Fibrillation: A Meta-analysis. Arch Med Res. 2015 Apr;46(3):199-206. doi: 10.1016/j.arcmed.2015.03.011. Epub 2015 May 14. PMID 25980945